CLINICAL TRIAL: NCT07186270
Title: Decoding the Interplay of Front-of-Pack Labels, Price, and Consumer Perceptions: Impact on Food Choices in Korea and Singapore
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Korea University (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Soye Shin, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 000273
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Consumer Behavior
Keywords: Front-of-pack labelling
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Intervention Model Description: At baseline, participants rate 8 menu items and 8 grocery items on a 5-point healthiness scale (1= least healthy, 5= healthiest) and their confidence. 6 menu items and 6 grocery items will be selected for experiment in study 1 and 2 respectively, prioritizing items with the largest perceived-actual healthiness gap, while ensuring varied confidence levels among items with similar gaps.
  Study 1: Participants read a hypothetical scenario about ordering meal for a co-worker. They will be randomized to 1 of the 4 conditions and asked to choose a menu item to order for their coworker.
  Study 2: Participants read a hypothetical cover story about a new brand Y of grocery item W and see pictures of different flavors with general health claim. They will be randomized to 1 of the 6 conditions. Participants indicate their likelihood of buying Brand Y in the hypothetical situation that they intend to purchase item W.
  Details of experiments in each study are discussed in the next section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study 1: Restaurant menu choice experiment (Experimental): Participants will read a hypothetical scenario about ordering a meal for a coworker. Participants will be told that their coworker has no dietary restrictions and is trying to eat healthier. They will be presented with two similar restaurant meal options, one priced higher than the other, with randomized assignments. In the label condition, a nutritional label for healthy foods, called the Healthy Choice Symbol adopted in Singapore, will be provided with an explanation of the labelling system. For both label and non-label conditions, participants will be asked to assess the healthfulness of each option using a standard 5-point scale (1-least healthy to 5-healthiest). Participants will then be asked to indicate which option to order for their coworker.
  Participants will be randomly assigned to one in four experimental arms.
  Interventions: Behavioral: Positively framed FOP labels (present versus absent) x Price (high versus low)
- Study 2: Grocery Food Item Choice Experiment (Experimental): Participants will read a hypothetical cover story about a new brand of a grocery item with generic health claims and see pictures of different flavors of this brand. Participants will be randomly assigned to either an average or a premium price condition and informed about the average price of other brands of the same item. They will be asked to indicate their perceived relative healthiness of the product compared to the products in other brands on a 5-point scale (1- least healthy to 5- healthiest). After assessment, they will see a high-grade label (grade A), low-grade label (grade D), or no label. For those exposed to labels, they will be given an explanation of the label and asked to indicate their perceived relative healthiness of the product again. In the end, all participants will indicate their intention to purchase items on a 7-point scale (1: least likely - 7: most likely).
  Participants will be assigned to one in six experimental arms.
  Interventions: Behavioral: Graded FOP labels (no label vs. high rating (grade A) vs. low rating (grade D)) x Price (average vs. premium)

INTERVENTIONS:
Behavioral: Positively framed FOP labels (present versus absent) x Price (high versus low) — The intervention combines either a front-of-pack (FOP) label that frames high nutrition or no FOP label with price variation. Products are randomly assigned to either receive a positively-framed FOP label or no label, and to either a high or a low price.
  This yields four experimental arms:
  1. Positively framed FOP label with high price
  2. Positively framed FOP label with low price
  3. No label with high price
  4. No label with low price
  Arms: Study 1: Restaurant menu choice experiment
Behavioral: Graded FOP labels (no label vs. high rating (grade A) vs. low rating (grade D)) x Price (average vs. premium) — The intervention combines either a graded front-of-pack (FOP) labelling or no FOP labelling with price variation. Products are randomly assigned to either receive a graded label or no label, and to either a premium or an average price.
  This yields six experimental arms:
  1. High grade (A) with premium price
  2. Low grade (D) with premium price
  3. No label with premium price
  4. High grade (A) with average price
  5. Low grade (D) with average price
  6. No label with average price
  Arms: Study 2: Grocery Food Item Choice Experiment

SUMMARY:
The global epidemic of obesity and chronic diseases has led to widespread use of front-of-package (FOP) nutrition labels. While existing research has established a link between FOP labels and consumer choices, the interplay between product types, consumer perceptions, and label effectiveness is underexplored. This study examines: 1) whether consumers perceive healthier food item as more expensive when healthiness is less obvious; 2) how FOP labels mediate the relationship among product characteristics, price, and consumer's belief about food healthiness and price on choices; and 3) whether food choice changes given a price, with and without FOP labels, are more prominent for products where the perceived healthiness by consumers significantly differs from label indications. The investigators will conduct experiments with online panelists in Korea and Singapore in two settings: restaurant menus and grocery items. Results will inform more impactful nutritional information policies for healthier food choices and improved population health.

DETAILED DESCRIPTION:
The investigators will conduct experiments in both Korea and Singapore, focusing on two settings with various food items: restaurant menu choices and grocery item selections. For each item, investigators will elicit consumers' prior belief about its healthiness. Our research builds upon the work of Haws et al. (2017), which demonstrated that US consumers tend to overgeneralize their belief about "expensive=healthy" to product categories where it is not true. This tendency potentially biases perceptions of healthy foods. The investigators aim to test this "expensive=healthy" intuition and its impact on food choice, with and without FOP labels, in Asian contexts. The investigators hypothesize that absent FOP labels, consumers will infer healthiness from price information (i.e., this product is expensive, so it must be healthy) and that providing FOP labels will reduce the reliance on this inference. The investigators also hypothesize that such effects of FOP labels are more prominent for products where the perceived healthiness by consumers significantly differs from the healthiness indicated by the labels. When the FOP labels show 'less healthy' for those expensive and perceived as 'healthy' products, consumers will update their prior belief about its healthiness and be more likely to drop the intuition 'expensive=healthiness' in decision-making and respond to a greater extent.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18-65 years residing in Korea
* Adults aged 21-65 years residing in Singapore

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Consumers behavior | Participants are expected to complete the online experiment in one sitting (within 24 hours). If they are disconnected from the survey platform, they are allowed up to two attempts to resume, with access to the platform disabled after 48 hours.
  Study 1: Participants achieve a response by choosing between two menu food items they would purchase for their co-worker in online experimental platform.
  Study 2: Participants rate their intention to purchase grocery items on a 7-point scale (1 = least likely, 7 = most likely) in online experimental platform.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyeon Lee, Principal Investigator — Korea University; Soye Shin, Principal Investigator — Duke-NUS Graduate Medical School